CLINICAL TRIAL: NCT01081730
Title: A Large US Health Insurance Claims Database Will be Used to Estimate the Incidence of Serious Outcomes in Patients With Psoriasis Treated With Ustekinumab and Other Types of Biological and Systemic Non-biological Treatments
Brief Title: Ustekinumab Safety and Surveillance Program Using the Ingenix NHI Database
Status: Completed | Type: Observational
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016723; CNTO1275PSO4006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis
Keywords: psoriasis; ustekinumab; anti-TNF biologics; non-anti-TNF biologics; systemic non-biological treatments
MeSH Terms: conditions — Psoriasis | interventions — Sociology; Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (5):
- 001: ustekinumab as prescribed
  Interventions: Biological: ustekinumab
- 002: anti-TNF biologics as prescribed
  Interventions: Biological: anti-TNF biologics
- 003: non-anti-TNF biologics as prescribed
  Interventions: Biological: non-anti-TNF biologics
- 004: systemic non-biological treatments as prescribed
  Interventions: Drug: systemic non-biological treatments
- 005: general population non-treated cohort
  Interventions: Other: general population

INTERVENTIONS:
Biological: anti-TNF biologics — as prescribed
  Groups: 002
Other: general population — non-treated cohort
  Groups: 005
Biological: non-anti-TNF biologics — as prescribed
  Groups: 003
Biological: ustekinumab — as prescribed
  Groups: 001
Drug: systemic non-biological treatments — as prescribed
  Groups: 004

SUMMARY:
The patients included in this observational study will be drawn from a research database containing claims and enrollment data for members of a large, geographically diverse US health plan. The objective of this study is to estimate the rate of serious infections, tuberculosis, malignancies, and other outcomes in psoriasis patients treated with ustekinumab, anti-tumor necrosis factor (TNF) biologics, non-anti-TNF biologics, or systemic non-biological treatments.

DETAILED DESCRIPTION:
The participants included in this study will be drawn from the Ingenix Normative Health Informatics Database, a proprietary research database containing claims and enrollment data dating back to 1993 for members of a large, geographically diverse US health plan. This study will include cohorts of participants who have claims consistent with a diagnosis of psoriasis and who initiate ustekinumab, anti-TNF biologics, non-anti-TNF biologics, or systemic non-biological treatments. Participants will be identified by claims bearing codes for dispensed drugs, procedures or diagnoses and followed after the launch of ustekinumab for up to 8 years. A sample of enrolled health plan members without claims evidence of diagnosis or treatment of psoriasis will also be selected. The claims database will be used to estimate the incidence of the primary outcomes of serious infections, tuberculosis (TB) and non-TB mycobacterial infections, malignancies such as lymphoma, and other selected outcomes. Potential cases of the study outcome identified through claims may be confirmed through medical record review. No study agents will be administered in this study. All patients will receive standard-of-care treatment as prescribed by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Complete medical coverage and pharmacy benefits
* Six months of continuous enrollment prior to the date of cohort entry

Exclusion Criteria:

* Participants will be excluded if they do not have information on age, gender or enrollment

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include cohorts of participants who have claims consistent with a diagnosis of psoriasis and who initiate ustekinumab, anti-TNF biologics, non-anti-TNF biologics, or systemic non-biological treatments
Sampling Method: Non-Probability Sample
Enrollment: 2040 (Actual)
Dates: Start 2010-02-09 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
To estimate the incidence of serious infections, tuberculosis and non-TB mycobacterial infections, malignancies, and other selected outcomes in patients with psoriasis initiating ustekinumab and other biological and systemic non-biological treatments | The study will be approximately 8 years in duration.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biologics Europe Clinical Trial, Study Director — Janssen Biotech, Inc.